CLINICAL TRIAL: NCT03118063
Title: Comparison of the Strength of Maximum Glute and Medium Glutenum Muscles Of Latin and Active Lombar Guidelines: A Clinical Test
Brief Title: Comparison of the Strength of Maximum Glute and Medium Glutenum Muscles Of Latin and Active Lombar Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Claudio Cazarini Junior, Physical therapist, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 62769916.6.0000.5479
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-02

CONDITIONS: Spinal Injuries; Low Back Pain
MeSH Terms: conditions — Spinal Injuries; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active trigger point (Experimental): Evaluation of the dynamometry of the maximum and medium gluteus muscles and correlate with the presence or not of trigger point
  Interventions: Diagnostic Test: Evaluation of pain by algometry
- Latent trigger point (Active Comparator): Assessment of the level of pain and function of asymptomatic individuals, compared with the time that they evolve with acute and chronic low back pain
  Interventions: Diagnostic Test: Evaluation of pain by algometry
- No trigger point (Active Comparator): Assessment of the level of pain and function of asymptomatic individuals, compared with the time that they evolve with acute and chronic low back pain
  Interventions: Diagnostic Test: Evaluation of pain by algometry

INTERVENTIONS:
Diagnostic Test: Evaluation of pain by algometry — Assessment of the level of pain and function of asymptomatic individuals, compared with the time that they evolve with acute and chronic low back pain

SUMMARY:
Contextualization: Trigger points are muscle nodules found in muscles. We can observe five different types of trigger point, in clinical practice two of them stand out, the active trigger point; Which is painful; And latent; Asymptomatic; Both of which are sensitive to palpation. Once the individual present these muscle nodules can develop pain and motor dysfunction. Studies indicate that the prevalence of trigger points is 95% of individuals with chronic musculoskeletal pain, but this prevalence is not yet clear in individuals with low back pain.

Objective: To compare the pain and function levels of patients with acute and chronic low back pain who, when asymptomatic, had trigger points compared to the pain and function levels of patients with acute and chronic low back pain who, when asymptomatic, had no trigger points.

Study design: Cohort study, two arms, blind evaluator, prospectively enrolled at baseline.

Location: This research will be conducted in the physiotherapy department at the Rehabilitation Center of the Brotherhood of Santa Casa de Misericórdia de São Paulo (ISCMSP).

Patients: 400 asymptomatic individuals Follow-up: Asymptomatic individuals will be assessed at baseline and over 3 years. You will be asked to contact the research department within 6 weeks of low back pain (acute) and after 12 weeks of low back pain (chronic). Participants will be allocated to two groups, trigger point group (n = 200) and group without trigger point (n = 200).

Outcomes: The pain intensity, function level and trigger point pain intensity outcomes will be evaluated at the baseline, within 6 weeks for the patient to present pain in the lumbar (acute) and after 12 weeks the pain persists (chronic)

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Age between 18 - 40 years;
* Asymptomatic;
* There is no treatment for lumbar spine, hip or knee.

Exclusion Criteria:

* Anterior lumbar spine surgeries;
* Severe spinal diseases (fracture, tumor, ankylosing spondylitis);
* Root conditions (herniated disc, spondylolisthesis);
* Congenital malformation;
* Pregnant women.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Function | 24 hours
  Evaluation of Function evaluation by the roland morris questionnaire
Pain scale | 24 hours
  Evaluation of pain by algometry

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil